CLINICAL TRIAL: NCT05473273
Title: Descriptive Analysis of Serum Immunological Markers During an Euploid Frozen Embryo Transfer in a Natural Cycle (NC).
Brief Title: Descriptive Analysis of Serum Immunological Markers During an Euploid Frozen Embryo Transfer in a Natural Cycle.
Status: Recruiting | Type: Observational
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Laura Marqueta Marques, Principal Investigator, ART Fertility Clinics LLC
Other Study IDs: 2206-ABU-004-LMM
Record Dates: First submitted 2022-07-22; First posted 2022-07-25 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: Infertility, Female
Keywords: infertilty; ivf; progesterone; estradiol; cytokines; immunology; Pharmacological effect of drugs; hormones
MeSH Terms: conditions — Infertility, Female; Long Qt Syndrome 3 | interventions — Progesterone; Estradiol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Natural Cycle Protocol: Ultrasound monitoring to monitor follicular and endometrial growth. Serial measurements of serum Lutenizing Hormone (LH), estradiol (E2), and progesterone (P4) to identify ovulation.
  Minimal endometrial thickness of 7 mm is required. No progesterone supplementation. Embryo transfer (ET) will be scheduled 5 days after the day of ovulation (120 hours of P4 exposure).
  Blood samples will be drawn to measure PIBF, IL-17, IFγ, IL-10, IL-4 and TGF-ß1 on day of ovulation (P4 rise), on the day before ET, on the day of ET and 3 and 10 days later, between 9 and 12 am.
  A blood test to measure beta human chorionic gonadotropin (ß-hCG) will be performed 3 and 10 days after ET and at 5 weeks +/- 3 days in case of pregnancy, between 9 and 12 am.
  In case of pregnancy, a blood test to measure PIBF, IL-17, IFγ, IL-10, IL-4 and TGF-ß1 will be performed at 5 weeks +/- 3 days between 9 and 12 am..
- Hormone Replacement Therapy Protocol: Ultrasound monitoring of endometrial growth and exclude growing follicle
  Oral Estradiol Valerate (Progyluton) 4 mg on cycle day 2 at 7 pm for 2 days. On 3rd day, increase dose to 6 mg. The dose may be increased based on endometrial thickness.
  Once endometrial thickness is at least 7 mm and trilaminar, after 10-15 days of Estradiol Valerate administration, start Endometrin 100 mg at 1 pm and 9 pm. From 2nd day onwards increase to 3 times daily. Continue Progyluton & Endometrin until 12 weeks of pregnancy
  ET on the 5th full day of Endometrin administration
  Blood test to measure PIBF, IL-17, IFγ, IL-4, IL-10 and TGF-ß1 on the 1st day of Endometrin supplementation (before 1st administration), on the 4th day of Endometrin administration, on the day of ET and 3 and10 days after, 4 to 7 hours after the morning administration.
  Blood test to measure beta human chorionic gonadotropin (ß-hCG) will be performed 3 and 10 days after ET and at 5 weeks +/- 3 days if pregnancy.
  Interventions: Drug: Endometrin 100Mg Vaginal Insert; Drug: Estradiol Valerate

INTERVENTIONS:
Drug: Endometrin 100Mg Vaginal Insert — Endometrin will start once endometrial thickness is equal or higher to 7 mm with a trilaminar appearance, after at least 10 days and always less than 16 days of estradiol administration. First day of supplementation a dose of 100mg will be administered at of at 1.pm and 9 pm. From the second day and onwards administration will be increased to three times daily, at 6 am, 2 pm and 10 pm
  Groups: Hormone Replacement Therapy Protocol
Drug: Estradiol Valerate — Estradiol valerate dose will be reduced to 4mg daily at 7 pm during the first two days of vaginal natural micronized progesterone supplementation and increased afterwards to 6 mg daily (2 mg at 10 am and 4 mg at 7 pm).
  Groups: Hormone Replacement Therapy Protocol

SUMMARY:
To describe the peripheral serum levels of the anti-inflammatory cytokines IL-4 (Interleukin-4), IL-10 (Interleukin-10), TGF-ß1 (Transforming Growth Factor beta1), the pro-inflammatory cytokines IL-17 (Interleukin-17), IFγ (Interferon Gamma) and the immune mediator PIBF (Progesterone-Induced Blocking Factor) along a single frozen euploid blastocyst transfer in a natural cycle (NC) or Hormone Replacement Therapy (HRT).

DETAILED DESCRIPTION:
This a prospective, observational study including 40 infertile patients undergoing a "single embryo transfer" (SET). Blood samples will be drawn for Progesterone-Induced Blocking Factor (PIBF), interleukin 17 (IL-17), Interferon Gamma (IFγ), Interleukin 10 (IL-10), Interleukin 4 (IL-4) and Transforming Growth Factor beta 1 (TGF-ß1) measurement on the day of ovulation in the natural cycle (NC) or first day of progesterone in the Hormone Replacement Therapy (HRT) protocol, on the day of embryo transfer (ET) and 3 and 10 days later, coinciding with the early and late embryo invasion stages respectively. In case of pregnancy, an additional blood test for PIBF, IL-17, IFγ, IL-10, IL-4, TGF-ß1 and ßHCG (Beta-Human Chorionic Gonadotropin) will be performed at 5 weeks +/- 3 days. The study will be performed at ART Fertility Clinics and the estimated completion time will be 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years to 40 years
* Having at least one good quality (grade A or B for inner mass cell and trophectoderm) day 5 or 6 chromosomally normal cryopreserved blastocyst available for transfer
* Single embryo transfer in a natural cycle (NC) or an Hormone Replacement Therapy (HRT) protocol
* Fresh ejaculate used for fertilization

Exclusion Criteria:

* Body mass index lower than 18.5 or equal or higher than 29 kg/m2
* Endometriosis or adenomyosis suspected by medical history (dysmenorrhea, dyspareunia, heavy or prolonged menstrual bleeding (> 8 days), chronic pelvic pain, catamenial rectal or bladder symptoms) or diagnosed by imaging (magnetic resonance imaging or ultrasonography)
* Uterine abnormalities
* Hydrosalpinx
* Insulin resistance or diabetes mellitus diagnosed by HbA1c 5.7 %
* Antiphospholipid syndrome
* Polycystic ovarian syndrome according to Rotterdam criteria: presence of at least two of the following: irregular cycles (< 21 or > 35 days or < 8 cycles a year), biochemical or clinical hyperandrogenism, ovarian ultrasound morphology (> 20 follicles per ovary on transvaginal scan) or Anti-mullerian hormone > 5,98 ng/ml
* History of recurrent miscarriage, defined as the loss of 2 or more pregnancies according to ESHRE guidelines
* History of implantation failure, considered as the lack of pregnancy after the transfer of 2 good-quality (grade A or B for inner mass cell and trophectoderm (29)) euploid embryos
* History or suspicion of Asherman syndrome
* Autoimmune disease
* Couple first degree consanguineous

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Infertile women undergoing a single frozen embryo transfer
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Blood levels of IL-4 (Interleukin 4) on the on the day of progesterone rise (NC) or first day of progesterone administration (HRT) | 1 day
  Blood levels of IL-4 on the on the day of progesterone rise (NC) or first day of progesterone administration (HRT)
Blood levels of IL-10 (Interleukin 10) on the on the day of progesterone rise (NC) or first day of progesterone administration (HRT) | 1 day
  Blood levels of IL-10 on the on the day of progesterone rise (NC) or first day of progesterone administration (HRT)
Blood levels of IL-17 (Interleukin 17) on the on the day of progesterone rise (NC) or first day of progesterone administration (HRT) | 1 day
  Blood levels of IL-17 on the on the day of progesterone rise (NC) or first day of progesterone administration (HRT)
Blood levels of TGF-ß1 (Transforming Growth Factor beta1) on the on the day of progesterone rise (NC) or first day of progesterone administration (HRT) | 1 day
  Blood levels of TGF-ß1 on the on the day of progesterone rise (NC) or first day of progesterone administration (HRT)
Blood levels of IFγ (Interferon gamma) on the on the day of progesterone rise (NC) or first day of progesterone administration (HRT) | 1 day
  Blood levels of IFγ on the on the day of progesterone rise (NC) or first day of progesterone administration (HRT)
Blood levels of PIBF on the on the day of progesterone rise (NC) or first day of progesterone administration (HRT) | 1 day
  Blood levels of PIBF on the on the day of progesterone rise (NC) or first day of progesterone administration (HRT)
Blood levels of IL-4 (Interleukin 4) on the day before embryo transfer | 1 day
  Blood levels of IL-4 on the day before embryo transfer
Blood levels of IL-10 (Interleukin 10) on the day before embryo transfer | 1 day
  Blood levels of IL-10 on the day before embryo transfer
Blood levels of IL-17 (Interleukin 17) on the day before embryo transfer | 1 day
  Blood levels of IL-17 on the day before embryo transfer
Blood levels of TGF-ß1 (Transforming Growth Factor beta1) on the day before embryo transfer | 1 day
  Blood levels of TGF-ß1 on the day before embryo transfer
Blood levels of IFγ (Interferon gamma) on the day before embryo transfer | 1 day
  Blood levels of IFγ on the day before embryo transfer
Blood levels of PIBF (Progesterone induced blocking factor) on the day before embryo transfer | 1 day
  Blood levels of PIBF on the day before embryo transfer
Blood levels of IL-4 (Interleukin 4) on the day of embryo transfer | 1 day
  Blood levels of IL-4 on the day of embryo transfer
Blood levels of IL-10 (Interleukin 10) on the day of embryo transfer | 1 day
  Blood levels of IL-10 on the day of embryo transfer
Blood levels of IL-17 (Interleukin 17) on the day of embryo transfer | 1 day
  Blood levels of IL-17 on the day of embryo transfer
Blood levels of TGF-ß1 (Transforming Growth Factor beta1) on the day of embryo transfer | 1 day
  Blood levels of TGF-ß1 on the day of embryo transfer
Blood levels of IFγ (Interferon gamma) on the day of embryo transfer | 1 day
  Blood levels of IFγ on the day of embryo transfer
Blood levels of PIBF (Progesterone induced blocking factor) on the day of embryo transfer | 1 day
  Blood levels of PIBF on the day of embryo transfer
Blood levels of IL-4 (Interleukin 4) three days after embryo transfer | 3 days
  Blood levels of IL-4 three days after embryo transfer
Blood levels of IL-10 (Interleukin 10) three days after embryo transfer | 3 days
  Blood levels of IL-10 three days after embryo transfer
Blood levels of IL-17 (Interleukin 17) three days after embryo transfer | 3 days
  Blood levels of IL-17 three days after embryo transfer
Blood levels of TGF-ß1 (Transforming Growth Factor beta1) three days after embryo transfer | 3 days
  Blood levels of TGF-ß1 three days after embryo transfer
Blood levels of IFγ (Interferon gamma) three days after embryo transfer | 3 days
  Blood levels of IFγ three days after embryo transfer
Blood levels of PIBF (Progesterone induced blocking factor) three days after embryo transfer | 3 days
  Blood levels of PIBF three days after embryo transfer
Blood levels of IL-4 (Interleukin 4) ten days after embryo transfer | 10 days
  Blood levels of IL-4 ten days after embryo transfer
Blood levels of IL-10 (Interleukin 10) ten days after embryo transfer | 10 days
  Blood levels of IL-10 ten days after embryo transfer
Blood levels of IL-17 (Interleukin 17) ten days after embryo transfer | 10 days
  Blood levels of IL-17 ten days after embryo transfer
Blood levels of TGF-ß1 (Transforming Growth Factor beta1) ten days after embryo transfer | 10 days
  Blood levels of TGF-ß1 ten days after embryo transfer
Blood levels of IFγ (Interferon gamma) ten days after embryo transfer | 10 days
  Blood levels of IFγ ten days after embryo transfer
Blood levels of PIBF (Progesterone induced blocking factor) ten days after embryo transfer | 10 days
  Blood levels of PIBF ten days after embryo transfer
Blood levels of IL-4 (Interleukin 4) in case of pregnancy at 5 weeks +/- 3 days | 5 weeks
  Blood levels of IL-4 in case of pregnancy at 5 weeks +/- 3 days
Blood levels of IL-10 (Interleukin 10) in case of pregnancy at 5 weeks +/- 3 days | 5 weeks
  Blood levels of IL-10 in case of pregnancy at 5 weeks +/- 3 days
Blood levels of IL-17 (Interleukin 17) in case of pregnancy at 5 weeks +/- 3 days | 5 weeks
  Blood levels of IL-17 in case of pregnancy at 5 weeks +/- 3 days
Blood levels of TGF-ß1 (Transforming Growth Factor beta1) in case of pregnancy at 5 weeks +/- 3 days | 5 weeks
  Blood levels of TGF-ß1 in case of pregnancy at 5 weeks +/- 3 days
Blood levels of IFγ (Interferon gamma) in case of pregnancy at 5 weeks +/- 3 days | 5 weeks
  Blood levels of IFγ in case of pregnancy at 5 weeks +/- 3 days
Blood levels of PIBF (Progesterone induced blocking factor) in case of pregnancy at 5 weeks +/- 3 days | 5 weeks
  Blood levels of PIBF in case of pregnancy at 5 weeks +/- 3 days
Blood levels of estradiol on the on the day of progesterone rise (NC) or first day of progesterone administration (HRT) | 1 day
  Blood levels of estradiol on the on the day of progesterone rise (NC) or first day of progesterone administration (HRT)
Blood levels of progesterone on the on the day of progesterone rise (NC) or first day of progesterone administration (HRT) | 1 day
  Blood levels of progesterone on the on the day of progesterone rise (NC) or first day of progesterone administration (HRT)
Blood levels of estradiol on the day before embryo transfer | 1 day
  Blood levels of estradiol on the day before embryo transfer
Blood levels of progesterone on the day before embryo transfer | 1 day
  Blood levels of progesterone on the day before embryo transfer
Blood levels of estradiol on the day of embryo transfer | 1 day
  Blood levels of estradiol on the day of embryo transfer
Blood levels of progesterone on the day of embryo transfer | 1 day
  Blood levels of progesterone on the day of embryo transfer
Blood levels of estradiol three days after embryo transfer | 3 days
  Blood levels of estradiol three days after embryo transfer
Blood levels of progesterone three days after embryo transfer | 3 days
  Blood levels of progesterone three days after embryo transfer
Blood levels of estradiol ten days after embryo transfer | 10 days
  Blood levels of estradiol ten days after embryo transfer
Blood levels of progesterone ten days after embryo transfer | 10 days
  Blood levels of progesterone ten days after embryo transfer
Blood levels of estradiol in case of pregnancy at 5 weeks +/- 3 days | 5 weeks
  Blood levels of estradiol in case of pregnancy at 5 weeks +/- 3 days
Blood levels of progesterone in case of pregnancy at 5 weeks +/- 3 days | 5 weeks
  Blood levels of progesterone in case of pregnancy at 5 weeks +/- 3 days
Blood levels of ß-hCG (Beta-Human Chorionic Gonadotropin) three days after embryo transfer | 3 days
  Blood levels of ß-hCG three days after embryo transfer
Blood levels of ß-hCG (Beta-Human Chorionic Gonadotropin) ten days after embryo transfer | 10 days
  Blood levels of ß-hCG ten days after embryo transfer
Blood levels of ß-hCG (Beta-Human Chorionic Gonadotropin) in case of pregnancy at 5 weeks +/- 3 days | 5 weeks
  Blood levels of ß-hCG in case of pregnancy at 5 weeks +/- 3 days

SECONDARY OUTCOMES:
Pregnancy rate | 10 days
  Number of patients with a ß-hCG > 5 IU out of the number of patients who underwent an embryo transfer.
Clinical pregnancy rate | 5 weeks and 3 days
  Number of patients with an ultrasonographic visible sac out of the number of patients who underwent an embryo transfer
Miscarriage rate | 12 weeks
  Number of patients with a pregnancy loss out of the number of patients who had a ß-hCG > 5 IU after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: LAURA MARQUETA MARQUES, Consultant, Principal Investigator — ART Fertility Clinics LLC
Locations (1):
- ART Fertility Clinics LLC, Abu Dhabi, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhang X, Wei H. Role of Decidual Natural Killer Cells in Human Pregnancy and Related Pregnancy Complications. Front Immunol. 2021 Aug 26;12:728291. doi: 10.3389/fimmu.2021.728291. eCollection 2021. PMID 34512661
- [Background] DeJong CS, Maurice NJ, McCartney SA, Prlic M. Human Tissue-Resident Memory T Cells in the Maternal-Fetal Interface. Lost Soldiers or Special Forces? Cells. 2020 Dec 16;9(12):2699. doi: 10.3390/cells9122699. PMID 33339211
- [Background] Diaz-Hernandez I, Alecsandru D, Garcia-Velasco JA, Dominguez F. Uterine natural killer cells: from foe to friend in reproduction. Hum Reprod Update. 2021 Jun 22;27(4):720-746. doi: 10.1093/humupd/dmaa062. PMID 33528013
- [Background] Lucas ES, Vrljicak P, Muter J, Diniz-da-Costa MM, Brighton PJ, Kong CS, Lipecki J, Fishwick KJ, Odendaal J, Ewington LJ, Quenby S, Ott S, Brosens JJ. Recurrent pregnancy loss is associated with a pro-senescent decidual response during the peri-implantation window. Commun Biol. 2020 Jan 21;3(1):37. doi: 10.1038/s42003-020-0763-1. PMID 31965050
- [Background] Lash GE, Robson SC, Bulmer JN. Review: Functional role of uterine natural killer (uNK) cells in human early pregnancy decidua. Placenta. 2010 Mar;31 Suppl:S87-92. doi: 10.1016/j.placenta.2009.12.022. Epub 2010 Jan 12. PMID 20061017
- [Background] Liu Y, Gao S, Zhao Y, Wang H, Pan Q, Shao Q. Decidual Natural Killer Cells: A Good Nanny at the Maternal-Fetal Interface During Early Pregnancy. Front Immunol. 2021 May 12;12:663660. doi: 10.3389/fimmu.2021.663660. eCollection 2021. PMID 34054831
- [Background] Robertson SA, Moldenhauer LM. Immunological determinants of implantation success. Int J Dev Biol. 2014;58(2-4):205-17. doi: 10.1387/ijdb.140096sr. PMID 25023687
- [Background] Mor G, Aldo P, Alvero AB. The unique immunological and microbial aspects of pregnancy. Nat Rev Immunol. 2017 Aug;17(8):469-482. doi: 10.1038/nri.2017.64. Epub 2017 Jun 19. PMID 28627518
- [Background] Piccinni MP, Raghupathy R, Saito S, Szekeres-Bartho J. Cytokines, Hormones and Cellular Regulatory Mechanisms Favoring Successful Reproduction. Front Immunol. 2021 Jul 28;12:717808. doi: 10.3389/fimmu.2021.717808. eCollection 2021. PMID 34394125
- [Background] AbdulHussain G, Azizieh F, Makhseed M, Raghupathy R. Effects of Progesterone, Dydrogesterone and Estrogen on the Production of Th1/Th2/Th17 Cytokines by Lymphocytes from Women with Recurrent Spontaneous Miscarriage. J Reprod Immunol. 2020 Aug;140:103132. doi: 10.1016/j.jri.2020.103132. Epub 2020 Apr 17. PMID 32380371
- [Background] Salem ML. Estrogen, a double-edged sword: modulation of TH1- and TH2-mediated inflammations by differential regulation of TH1/TH2 cytokine production. Curr Drug Targets Inflamm Allergy. 2004 Mar;3(1):97-104. doi: 10.2174/1568010043483944. PMID 15032646
- [Background] Szekeres-Bartho J. The Role of Progesterone in Feto-Maternal Immunological Cross Talk. Med Princ Pract. 2018;27(4):301-307. doi: 10.1159/000491576. Epub 2018 Jun 27. PMID 29949797
- [Background] Wang W, Sung N, Gilman-Sachs A, Kwak-Kim J. T Helper (Th) Cell Profiles in Pregnancy and Recurrent Pregnancy Losses: Th1/Th2/Th9/Th17/Th22/Tfh Cells. Front Immunol. 2020 Aug 18;11:2025. doi: 10.3389/fimmu.2020.02025. eCollection 2020. PMID 32973809
- [Background] Raghupathy R, Szekeres-Bartho J. Progesterone: A Unique Hormone with Immunomodulatory Roles in Pregnancy. Int J Mol Sci. 2022 Jan 25;23(3):1333. doi: 10.3390/ijms23031333. PMID 35163255
- [Background] Zhao Y, Zhang T, Guo X, Wong CK, Chen X, Chan YL, Wang CC, Laird S, Li TC. Successful implantation is associated with a transient increase in serum pro-inflammatory cytokine profile followed by a switch to anti-inflammatory cytokine profile prior to confirmation of pregnancy. Fertil Steril. 2021 Apr;115(4):1044-1053. doi: 10.1016/j.fertnstert.2020.10.031. Epub 2020 Nov 30. PMID 33272613
- [Background] Murphy SP, Tayade C, Ashkar AA, Hatta K, Zhang J, Croy BA. Interferon gamma in successful pregnancies. Biol Reprod. 2009 May;80(5):848-59. doi: 10.1095/biolreprod.108.073353. Epub 2009 Jan 21. PMID 19164174
- [Background] Chaouat G, Menu E, Clark DA, Dy M, Minkowski M, Wegmann TG. Control of fetal survival in CBA x DBA/2 mice by lymphokine therapy. J Reprod Fertil. 1990 Jul;89(2):447-58. doi: 10.1530/jrf.0.0890447. PMID 2119428
- [Background] Xu WM, Xiao ZN, Wang XB, Huang Y. IL-17 Induces Fetal Loss in a CBA/JxBALB/c Mouse Model, and an Anti-IL-17 Antibody Prevents Fetal Loss in a CBA/JxDBA/2 Mouse Model. Am J Reprod Immunol. 2016 Jan;75(1):51-8. doi: 10.1111/aji.12437. Epub 2015 Oct 17. PMID 26474535
- [Background] Kao LC, Tulac S, Lobo S, Imani B, Yang JP, Germeyer A, Osteen K, Taylor RN, Lessey BA, Giudice LC. Global gene profiling in human endometrium during the window of implantation. Endocrinology. 2002 Jun;143(6):2119-38. doi: 10.1210/endo.143.6.8885. PMID 12021176
- [Background] Wu HX, Jin LP, Xu B, Liang SS, Li DJ. Decidual stromal cells recruit Th17 cells into decidua to promote proliferation and invasion of human trophoblast cells by secreting IL-17. Cell Mol Immunol. 2014 May;11(3):253-62. doi: 10.1038/cmi.2013.67. Epub 2014 Mar 17. PMID 24633013
- [Background] Yang D, Dai F, Yuan M, Zheng Y, Liu S, Deng Z, Tan W, Chen L, Zhang Q, Zhao X, Cheng Y. Role of Transforming Growth Factor-beta1 in Regulating Fetal-Maternal Immune Tolerance in Normal and Pathological Pregnancy. Front Immunol. 2021 Aug 31;12:689181. doi: 10.3389/fimmu.2021.689181. eCollection 2021. PMID 34531852
- [Background] Keskin DB, Allan DS, Rybalov B, Andzelm MM, Stern JN, Kopcow HD, Koopman LA, Strominger JL. TGFbeta promotes conversion of CD16+ peripheral blood NK cells into CD16- NK cells with similarities to decidual NK cells. Proc Natl Acad Sci U S A. 2007 Feb 27;104(9):3378-83. doi: 10.1073/pnas.0611098104. Epub 2007 Feb 20. PMID 17360654
- [Background] Matalka KZ. The effect of estradiol, but not progesterone, on the production of cytokines in stimulated whole blood, is concentration-dependent. Neuro Endocrinol Lett. 2003 Jun-Aug;24(3-4):185-91. PMID 14523355
- [Background] Bourdon M, Santulli P, Jeljeli M, Vannuccini S, Marcellin L, Doridot L, Petraglia F, Batteux F, Chapron C. Immunological changes associated with adenomyosis: a systematic review. Hum Reprod Update. 2021 Jan 4;27(1):108-129. doi: 10.1093/humupd/dmaa038. PMID 33099635
- [Background] Conrad KP, Baker VL. Corpus luteal contribution to maternal pregnancy physiology and outcomes in assisted reproductive technologies. Am J Physiol Regul Integr Comp Physiol. 2013 Jan 15;304(2):R69-72. doi: 10.1152/ajpregu.00239.2012. Epub 2012 Oct 24. PMID 23100030
- [Background] Chen JZ, Sheehan PM, Brennecke SP, Keogh RJ. Vessel remodelling, pregnancy hormones and extravillous trophoblast function. Mol Cell Endocrinol. 2012 Feb 26;349(2):138-44. doi: 10.1016/j.mce.2011.10.014. Epub 2011 Oct 25. PMID 22051447
- [Background] Labarta E, Mariani G, Paolelli S, Rodriguez-Varela C, Vidal C, Giles J, Bellver J, Cruz F, Marzal A, Celada P, Olmo I, Alama P, Remohi J, Bosch E. Impact of low serum progesterone levels on the day of embryo transfer on pregnancy outcome: a prospective cohort study in artificial cycles with vaginal progesterone. Hum Reprod. 2021 Feb 18;36(3):683-692. doi: 10.1093/humrep/deaa322. PMID 33340402
- [Background] Labarta E, Sebastian-Leon P, Devesa-Peiro A, Celada P, Vidal C, Giles J, Rodriguez-Varela C, Bosch E, Diaz-Gimeno P. Analysis of serum and endometrial progesterone in determining endometrial receptivity. Hum Reprod. 2021 Oct 18;36(11):2861-2870. doi: 10.1093/humrep/deab184. PMID 34382075
- [Background] Abdala A, Elkhatib I, Bayram A, Arnanz A, El-Damen A, Melado L, Lawrenz B, Fatemi HM, De Munck N. Day 5 vs day 6 single euploid blastocyst frozen embryo transfers: which variables do have an impact on the clinical pregnancy rates? J Assist Reprod Genet. 2022 Feb;39(2):379-388. doi: 10.1007/s10815-021-02380-1. Epub 2022 Jan 22. PMID 35064434
- [Background] Munro MG, Critchley HOD, Fraser IS; FIGO Menstrual Disorders Committee. The two FIGO systems for normal and abnormal uterine bleeding symptoms and classification of causes of abnormal uterine bleeding in the reproductive years: 2018 revisions. Int J Gynaecol Obstet. 2018 Dec;143(3):393-408. doi: 10.1002/ijgo.12666. Epub 2018 Oct 10. PMID 30198563
- [Background] Rotterdam ESHRE/ASRM-Sponsored PCOS Consensus Workshop Group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome. Fertil Steril. 2004 Jan;81(1):19-25. doi: 10.1016/j.fertnstert.2003.10.004. PMID 14711538
- [Background] Calzada M, Lopez N, Noguera JA, Mendiola J, Hernandez AI, Corbalan S, Sanchez M, Torres AM. AMH in combination with SHBG for the diagnosis of polycystic ovary syndrome. J Obstet Gynaecol. 2019 Nov;39(8):1130-1136. doi: 10.1080/01443615.2019.1587604. Epub 2019 Jun 17. PMID 31208261
- [Background] Fatemi HM, Kyrou D, Bourgain C, Van den Abbeel E, Griesinger G, Devroey P. Cryopreserved-thawed human embryo transfer: spontaneous natural cycle is superior to human chorionic gonadotropin-induced natural cycle. Fertil Steril. 2010 Nov;94(6):2054-8. doi: 10.1016/j.fertnstert.2009.11.036. Epub 2010 Jan 25. PMID 20097333